CLINICAL TRIAL: NCT03206697
Title: Definition: Evaluation of Mitichondrial Values and it Relationship With Embryo Metabolism and Mitochondrial Homeostasis.
Brief Title: mtDNA and Embryo Metabolism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Collaborators: Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: 1606-VLC-047-MD
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Embryo Metabolic Activity
Keywords: mitochondrial copy, number and energy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aneuploid mitochondria: Mitochondrial DNA content and metabolic parameters
  Interventions: Other: Mitochondrial DNA content and metabolic parameters

INTERVENTIONS:
Other: Mitochondrial DNA content and metabolic parameters — Analyze the correlation between the mitochondrial DNA content and metabolic parameters.

SUMMARY:
The present study has the objective to study whether the mitochondrial DNA copy number values that can be generated when human embryos are analyzed for chromosomal content before embryo transfer correlates with the actual number of mitochondria as well as their energy requirements of the human embryo.

DETAILED DESCRIPTION:
The possibility of analyzing trophectoderm cells from human blastocyst during preimplantational genetic testing offers the opportunity of analyzing not only the chromosomal constitution of the trophoblastic cells, and by extension, to infer not with certain degree of uncertainty, the chromosomal content in the inner cell cells mass and the entire embryo; but analyzing other interesting aspects related to cellular physiology such us the mtDNA content.

The number of mitochondrial copy number has a huge variation among oocytes from the same cohort and also from oocytes from different patients. It is believed that this initial number of mtDNA content is correlated with the ability of oocytes to fertilized and to achieve blastocyst stage. Whatever the initial concentration of mtDNA a given oocyte will have, it expected to equally segregate into the number of blastomeres along embryo development, so the mtDNA copy number of per daughter cell will transiently decrease, being the smallest at the blastocyst stage. Studies in different mammalian species including humans have shown that mtDNA replication does not occur before morula stage so the mitochondrial content of the oocytes should be enough to sustain embryo development before implantation occurs.

The net amount of mitochondrial DNA will exponentially increase at blastocyst stage coinciding with an increases in oxygen consumption. Despite the mtDNA copy number is higher in ICM compared to TE cells the proportion of moderate and high activity mitochondria is higher in the TE cells. This also agrees with mitochondrial morphological changes in the trophectoderm cells where mitochondria are much more elongated, less matrix electrodense and have more cristae, in ICM the will be rounded and more electrodense.

The objective of the present work is to analyze whether a correlation exist between the mitochondrial DNA copy number and both the actual number of mitochondria in the blastocyst and the metabolic needs of the human blastocysts and the ATP production.

ELIGIBILITY:
Inclusion Criteria of women whose blastocysts will undergo PGT-A and be eligible for study:

* > 38 years old
* Sperm count: > 2 million spermatozoids/ml
* Oocytes retrieved > 4 oocytes MII
* Antral Follicles (AFC: ≥4)

Ages: 5 Days to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Blastocysts from women undergoing PGT-A and available for analysis )
Sampling Method: Probability Sample
Enrollment: 171 (Estimated)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Correlation between mitochondrial DNA content and number of mitochondria and Correlation between mitochondrial DNA content and metabolic turnover | Each embryo will need an average of one week for assessment
  Correlation index between each variable

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Jose DeLosSantos, Valencia, Spain